CLINICAL TRIAL: NCT00003020
Title: Protocol for a Phase I Study of Intrathecal LMB-7 (Single-Chain Immunotoxin Constructed From Monoclonal Antibody B3-Pseudomonas Exotoxin PE 38) [IND 5863, NSC 658931] in the Treatment of Patients With Leptomeningeal Neoplasms
Brief Title: LMB-7 Immunotoxin in Treating Patients With Leptomeningeal Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000065605; DUMC-0511-99-3R2; DUMC-000428-00-3R3; DUMC-424-98-3R1; DUMC-460-97-3; NCI-T96-0012
Record Dates: First submitted 1999-11-01; First posted 2004-05-19 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: leptomeningeal metastases
MeSH Terms: conditions — Central Nervous System Neoplasms; Meningeal Carcinomatosis | interventions — immunotoxin LMB-7

INTERVENTIONS:
Biological: LMB-7 immunotoxin

SUMMARY:
RATIONALE: LMB-7 immunotoxin can locate tumor cells and kill them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of LMB-7 immunotoxin in treating patients who have leptomeningeal metastases metastases.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity of intrathecal LMB-7 immunotoxin in patients with leptomeningeal metastases. II. Identify objective therapeutic responses in this group of patients.

OUTLINE: This is a dose escalation study. Patients receive LMB-7 intrathecally on days 1, 3, and 5. Treatment may be repeated every 4 weeks if the patient does not demonstrate HAMA neutralizing antibodies to PE-38 in CSF, has stable or responding disease, and has not experienced greater than grade II toxicity. Three to six patients are entered at each dose level. Dose escalation continues until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience grade 3 or worse toxicity or a neuroradiology toxicity score of 10 or greater.

PROJECTED ACCRUAL: Approximately 15 to 24 patients will be accrued over one year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven primary intracranial or extraneural neoplasm with leptomeningeal metastases At least 30% of malignant cells in the cerebrospinal fluid, primary tumor, or metastatic tumor must react with the B3 mouse monoclonal antibody

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 50-100% Life expectancy: Not specified Hematopoietic: ANC greater than 1000/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin less than 1.5 mg/dL Renal: Creatinine less than 1.2 mg/dL Pulmonary: DLCO at least 60 Other: No neutralizing antibodies to Pseudomonas exotoxin Not pregnant or nursing Not allergic to penicillin

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No chemotherapy within past 4 weeks (6 weeks for nitrosoureas) unless there is evidence of disease progression in CNS No concurrent chemotherapy Endocrine therapy: Patients receiving corticosteroids must be on stable dose for 10 days prior to entry Radiotherapy: No radiotherapy to disease site within past 3 months unless there is evidence of disease progression in CNS No concurrent radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 1997-09; Primary Completion 2000-09 (Actual); Study Completion 2000-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darell D. Bigner, MD, PhD, Study Chair — Duke Cancer Institute
Locations (2):
- United States (2):
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania